CLINICAL TRIAL: NCT05569785
Title: Exploring the Short-Term Effect of Bariatric Surgery on Muscle Structure And Function; Followed By A Feasibility Assessment Of Exercise Intervention Post Bariatric Surgery
Brief Title: Bariatric Surgery and Exercise Interventions: Effects on Muscle
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 22012
Record Dates: First submitted 2022-05-30; First posted 2022-10-06 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Bariatric Surgery Candidate; Obesity
Keywords: resistance exercise therapy
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: A single-centre feasibility research programme
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 Resistance Exercise Therapy Feasibility (Active Comparator): One group who have been randomised to receive 4 weeks of Resistance Exercise Therapy to explore the feasibility of introducing such a programme in the bariatric population.
  Interventions: Other: Resistance Exercise Therapy
- Group 2 Standard Care (No Intervention): This group have been randomised to receive standard care post surgery.

INTERVENTIONS:
Other: Resistance Exercise Therapy — 4 weeks of Resistance Exercise Therapy. This is a 4 week resistance exercise training programme that can be completed at home. The programme is designed to be progressive. It was designed by a bariatric physiotherapist and an exercise physiologist. This exercise programme will be discussed at the screening visit, educational material will be provided to the participants who are randomised to the intervention RET group.
  Safety advice will be given to each eligible participant to ensure that if they feel unwell, develop chest pain/tightness, then they must seek advice from GP/urgent care if necessary. The exercises will need to be performed at least three times a week. Compliance will be monitored with Fitbit downloads at each visit. Fitbits will be worn during exercise sessions only.
  Arms: Group 1 Resistance Exercise Therapy Feasibility

SUMMARY:
The purpose of this project is to assess the effects of bariatric surgery on muscle structure and function as well as investigating the feasibility of undertaking an exercise intervention post-surgery.

DETAILED DESCRIPTION:
A single-centre feasibility research programme based at the Royal Derby Hospital centre of the University of Nottingham. This is an exploratory and feasibility study. Muscle structure and function of 12 patients will be assessed before bariatric surgery and at 6 weeks, and then 10 weeks, after surgery. After 6 weeks, participants will be randomised into two groups. Group 1 will undergo a 4 week Resistance Exercise Training (RET). Group 2 will undergo standard care procedure. The total duration of programme we are aiming for is 13-14 weeks prior to bariatric surgery and exercise intervention for 4 weeks after bariatric surgery.

ELIGIBILITY:
Inclusion Criteria:

* Obese adults (BMI greater than or equal to 35 kg/m2)
* Age range 18-70 years old
* Scheduled for RYGB surgery or sleeve gastrectomy surgery.
* Ability to give informed consent

Exclusion Criteria:

* Patients who are not fit or not suitable for RYGB or Sleeve Gastrectomy as per Tier 4 Bariatric Surgery MDT.
* For those high-risk patients who are fast tracked to surgery, we will exclude patients with a NYHA >3 or 4 heart failure status and those with end stage renal failure.
* BMI greater than or equal to 60

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
To assess the effects of bariatric surgery on skeletal muscle ultrasound thickness. | Total duration of study per participant is expected to be 13 to 14 weeks
  This will be assessed using muscle ultrasound and units (mm)
To assess the effects of bariatric surgery on skeletal muscle cross sectional area (cm2) | Total duration of study per participant is expected to be 13 to 14 weeks
  This will be assessed using muscle ultrasound
Assessment of percentage of patients who were retained throughout the intervention arm of the study | Total duration of study per participant is expected to be 13 to 14 weeks
  To be measured as percentage.
Assessment of percentage of patients who were compliant with the intervention arm of the study. To be guided by FitBit monitor use. | Total duration of study per participant is expected to be 13 to 14 weeks
  This assessment will be measured as percentage of patients who met compliance targets with the intervention arm for the study.
Assessment of number of patients who were recruited to the study | Total duration of study per participant is expected to be 13 to 14 weeks
  This assessment will be measured as a simple numeric value

SECONDARY OUTCOMES:
Fasting glucose | Total duration of study per participant is expected to be 13 to 14 weeks, there will be bloods taken on each in-person study day. Plan is for 3 of these days, screening bloods will be reviewed from the NHS interface.
  These results will be undertaken by analysing blood samples taken by venepuncture of participants. Units will be mmol .
Skeletal muscle architecture (fibre length) | Total duration of study per participant is expected to be 13 to 14 weeks, ultrasounds will be performed at each in-person study day. performed on each in-person study day
  An ultrasound scan will be used for the purpose of this measurement. Units (mm).
Muscle fatigability (maximum voluntary contractions) | Total duration of study per participant is expected to be 13 to 14 weeks, each assessment for this outcome will take place at the in-person study days.
  This is the maximal force-generating capacity of a muscle or group of muscles
Lean body mass using BIA and D3 creatine | Total duration of study per participant is expected to be 13 to 14 weeks, each participant will be provided with the resources to facilitate these assessments at their in-person study days, urine collections will be returned later..
  These are stable biomarkers that have been previously used in research. It acts in the body as creatine, which is a naturally occurring substance.
Motor control in force tracking | Total duration of study per participant is expected to be 13 to 14 weeks, these assessments will be performed at each in-person study day.
  As part of the Short Physical Performance Battery Test
Balance using the Timed Up and Go (TUG) test | Total duration of study per participant is expected to be 13 to 14 weeks, these assessments will be performed at each in-person study day.
  As part of the Short Physical Performance Battery Test
Balance in Gait and Motion testing | Total duration of study per participant is expected to be 13 to 14 weeks, these assessments will be performed at each in-person study day.
  As part of the Short Physical Performance Battery Test
Hand grip strength | Total duration of study per participant is expected to be 13 to 14 weeks, these assessments will be performed at each in-person study day.
  The purpose of the handgrip strength test is to measure the maximum isometric strength of the hand and forearm muscles
Predicted maximum oxygen consumption (VO2 max) in step box test | Total duration of study per participant is expected to be 13 to 14 weeks, these assessments will be performed at each in-person study day.
  As part of the Short Physical Performance Battery Test
Skin fold and body circumference measurements | Total duration of study per participant is expected to be 13 to 14 weeks, these assessments will be performed at each in-person study day.
  To assess for any interval change
Quality of life measurements using IPAQ questionnaire | Total duration of study per participant is expected to be 13 to 14 weeks, these assessments will be performed at each in-person study day.
  Questionnaires are performed to standardise the assessment of quality of life from the patient perspective. IPAQ questionnaire contains open-ended questions surrounding individuals' last 7-day recall of physical activity
insulin resistance (HOMA-IR) | Total duration of study per participant is expected to be 13 to 14 weeks, these assessments will be performed at each in-person study day.
  These results will be undertaken by analysing blood samples taken by venepuncture of participants. Units will be nmol/L.
Skeletal muscle architecture (pennation angle) | Total duration of study per participant is expected to be 13 to 14 weeks, these assessments will be performed at each in-person study day.
  An ultrasound scan will be used for the purpose of this measurement, units will be in degrees.
Quality of life measurements using SF-36 questionnaire | Total duration of study per participant is expected to be 13 to 14 weeks, these assessments will be performed at each in-person study day.
  Questionnaires are performed to standardise the assessment of quality of life from the patient perspective.This questionnaire uses a likert scale as means of assessment.

CONTACTS AND LOCATIONS:
Locations (1):
- COMAP, Derby, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No plan to do so

REFERENCES:
- [Background] Wadstrom C, Backman L, Forsberg AM, Nilsson E, Hultman E, Reizenstein P, Ekman M. Body composition and muscle constituents during weight loss: studies in obese patients following gastroplasty. Obes Surg. 2000 Jun;10(3):203-13. doi: 10.1381/096089200321643313. PMID 10932257
- [Background] Alba DL, Wu L, Cawthon PM, Mulligan K, Lang T, Patel S, King NJ, Carter JT, Rogers SJ, Posselt AM, Stewart L, Shoback DM, Schafer AL. Changes in Lean Mass, Absolute and Relative Muscle Strength, and Physical Performance After Gastric Bypass Surgery. J Clin Endocrinol Metab. 2019 Mar 1;104(3):711-720. doi: 10.1210/jc.2018-00952. PMID 30657952
- [Background] Haeffener MP, Ferreira GM, Barreto SS, Arena R, Dall'Ago P. Incentive spirometry with expiratory positive airway pressure reduces pulmonary complications, improves pulmonary function and 6-minute walk distance in patients undergoing coronary artery bypass graft surgery. Am Heart J. 2008 Nov;156(5):900.e1-900.e8. doi: 10.1016/j.ahj.2008.08.006. Epub 2008 Oct 5. PMID 19061704
- [Background] Li C, Carli F, Lee L, Charlebois P, Stein B, Liberman AS, Kaneva P, Augustin B, Wongyingsinn M, Gamsa A, Kim DJ, Vassiliou MC, Feldman LS. Impact of a trimodal prehabilitation program on functional recovery after colorectal cancer surgery: a pilot study. Surg Endosc. 2013 Apr;27(4):1072-82. doi: 10.1007/s00464-012-2560-5. Epub 2012 Oct 9. PMID 23052535
- [Background] Santa Mina D, Clarke H, Ritvo P, Leung YW, Matthew AG, Katz J, Trachtenberg J, Alibhai SM. Effect of total-body prehabilitation on postoperative outcomes: a systematic review and meta-analysis. Physiotherapy. 2014 Sep;100(3):196-207. doi: 10.1016/j.physio.2013.08.008. Epub 2013 Nov 13. PMID 24439570
- [Background] Herring LY, Stevinson C, Carter P, Biddle SJH, Bowrey D, Sutton C, Davies MJ. The effects of supervised exercise training 12-24 months after bariatric surgery on physical function and body composition: a randomised controlled trial. Int J Obes (Lond). 2017 Jun;41(6):909-916. doi: 10.1038/ijo.2017.60. Epub 2017 Mar 6. PMID 28262676